CLINICAL TRIAL: NCT02579239
Title: An Open-Label, Intrapatient Dose Escalation Study to Evaluate the Safety, Tolerability, Immunogenicity, and Biological Activity of ATYR1940 in Patients With Limb Girdle and Facioscapulohumeral Muscular Dystrophies
Brief Title: Evaluate Safety and Biological Activity of ATYR1940 in Participants With Limb Girdle Muscular Dystrophy 2B (LGMD2B) and Facioscapulohumeral Muscular Dystrophy (FSHD)
Acronym: FSHD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: aTyr Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATYR1940-C-004; 2015-001910-88 (EudraCT Number)
Record Dates: First submitted 2015-09-28; First posted 2015-10-19 (Estimated); Results first posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-09

CONDITIONS: Limb-Girdle Muscular Dystrophies; Facioscapulohumeral Muscular Dystrophy
Keywords: LGMD2B; FSHD
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle; Muscular Dystrophy, Facioscapulohumeral; Limb-girdle muscular dystrophy, type 2B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A - FSHD (Experimental): Participants with FSHD will receive single dose of placebo intravenous (IV) infusion followed by ATYR1940 IV infusion at doses of 0.3 up to 1.0 milligrams/kilograms (mg/kg) once weekly for 8 weeks and then twice weekly for 4 weeks using intraparticipant dose escalation for up to 12 weeks.
  Interventions: Biological: ATYR1940; Biological: Placebo
- Group B - LGMD2B and FSHD (Experimental): Participants with LGMD2B and FSHD will receive single dose of placebo IV infusion followed by ATYR1940 IV infusion at doses of 0.3 up to 1.0 and 3.0 mg/kg once weekly for 8 weeks and then twice weekly for 4 weeks using intraparticipant dose escalation for up to 12 weeks.
  Interventions: Biological: ATYR1940; Biological: Placebo

INTERVENTIONS:
Biological: ATYR1940 — Concentrate for solution for infusion
Biological: Placebo — Concentrate for solution for infusion

SUMMARY:
The purpose of this study is to assess the safety and biological activity of ATYR1940 in participants with LGMD2B and FSHD.

ELIGIBILITY:
Inclusion Criteria:

* Provided informed consent.
* Investigator's opinion, participant is willing and able to complete all study procedures and comply with the study visit schedule.

Participant with LGMD2B:

* Established, genetically confirmed diagnosis of LGMD2B.
* Either the presence of a short tau inversion recovery (STIR) positive muscle on lower extremity skeletal muscle magnetic resonance imaging (MRI), or, if no STIR positive muscles, meets muscle biomarker criteria.

Participant with FSHD:

* Established, genetically confirmed diagnosis of FSHD.
* The presence of a STIR positive muscle on lower extremity skeletal muscle MRI.

Exclusion Criteria:

* Currently receiving treatment with an immunomodulatory agent, including targeted biological therapies within the 3 months before baseline; corticosteroids within 3 months before baseline; or high-dose non-steroidal anti-inflammatory agents within 2 weeks before baseline.
* Currently receiving curcumin or albuterol; use of a product that putatively enhances muscle growth on a chronic basis within 30 days before baseline; statin treatment initiation or significant adjustment to statin regimen within 3 months before baseline (stable, chronic statin use is permissible).
* Use of an investigational product or device within 30 days before baseline.
* Evidence of an alternative diagnosis other than LGMD2B or FSHD or a coexisting myopathy or dystrophy, based on prior muscle biopsy or other available investigations.
* History of severe restrictive or obstructive lung disease or evidence for interstitial lung disease on screening chest radiograph.
* History of anti-synthetase syndrome, prior Jo-1 Ab-positivity, or a positive or equivocally positive Jo-1 Ab test result during screening.
* Chronic infection, such as hepatitis B, hepatitis C, or human immunodeficiency virus or a history of tuberculosis.
* Vaccination within 8 weeks before baseline or vaccination is planned during study participation.
* Symptomatic cardiomyopathy or severe cardiac arrhythmia that may in the Investigator's opinion, limit the participant's ability to complete the study protocol.
* Muscle biopsy within 30 days before baseline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2016-10-05 (Actual); Study Completion 2016-10-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - University of California, Irvine, ALS and Neuromuscular Center, Irvine, California
  - Kennedy Krieger Institute; The Johns Hopkins University School of Medicine, Baltimore, Maryland
  - OSU Wexner Medical Center, Columbus, Ohio
- Rigshospitalet, University of Copenhagen, Copenhagen, Denmark
- France (2):
  - Centre d'nvestigation Clinique - Centre de Pharmacologie Clinique et d'Evaluations Thérapeutiques (CICCPCET), Marseille
  - Institut de Myologie, Hôpital Pitié-Salpêtrière, Paris

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A - FSHD: Participants with FSHD received single dose of placebo intravenous (IV) infusion followed by ATYR1940 IV infusion at doses of 0.3 up to 1.0 milligrams/kilograms (mg/kg) once weekly for 8 weeks and then twice weekly for 4 weeks using intraparticipant dose escalation for up to 12 weeks.
- Group B - LGMD2B and FSHD: Participants with LGMD2B and FSHD received single dose of placebo IV infusion followed by ATYR1940 IV infusion at doses of 0.3 up to 1.0 and 3.0 mg/kg once weekly for 8 weeks and then twice weekly for 4 weeks using intraparticipant dose escalation for up to 12 weeks.
Period: Overall Study
Arm/Group | Group A - FSHD | Group B - LGMD2B and FSHD
Started | 4 | 14
Received at Least 1 Dose of Study Drug | 4 | 14
Completed | 4 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 full or partial dose of ATYR1940 and had a post-infusion safety observation.
Groups:
- Group A - FSHD: Participants with FSHD received single dose of placebo IV infusion followed by ATYR1940 IV infusion at doses of 0.3 up to 1.0 mg/kg once weekly for 8 weeks and then twice weekly for 4 weeks using intraparticipant dose escalation for up to 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Group A - FSHD | Group B - LGMD2B and FSHD | Total
Number analyzed (Participants) | 4 | 14 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 14 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (4.97) | 36.3 (11.15) | 38.2 (10.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 8
  Male | 3 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAEs were defined as adverse events (AEs) with an onset following administration of the first dose of study drug. An AE was defined as any untoward medical occurrence in a participant administered study drug and that does not necessarily have a causal relationship with the study drug. Worsening of a pre-existing medical condition should have been considered an AE if there was either an increase in severity, frequency, or duration of the condition or an association with significantly worse outcomes. An SAE was defined as any AE that, in the view of either the Investigator or Sponsor, resulted in any of the following outcomes as fatal, life-threatening, required in-participant hospitalization or prolongation of existing hospitalization, in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or an important medical event. A summary of all SAEs and Other AEs (nonserious) regardless of causality is located in 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (up to Week 25)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - FSHD | Group B - LGMD2B and FSHD
Number analyzed (Participants) | 4 | 14
Participants
  TEAEs | 4 | 14
  SAEs | 0 | 0

2. Primary Outcome: Number of Participants With a Clinically Significant Electrocardiogram (ECG) Abnormality Leading to a TEAE
Description: ECG parameters that were evaluated included heart rate, PR, and QR and QT intervals. A clinically significant ECG abnormality was based upon the Investigator's discretion. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (up to Week 25)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - FSHD | Group B - LGMD2B and FSHD
Number analyzed (Participants) | 4 | 14
Participants | 0 | 0

3. Primary Outcome: Number of Participants With a Clinically Significant Pulmonary Function Event Resulting in a TEAE
Description: Pulmonary evaluations included pulmonary function tests and pulse oximetry. Clinically significant changes were to be reported as adverse events. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (up to Week 25)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - FSHD | Group B - LGMD2B and FSHD
Number analyzed (Participants) | 4 | 14
Participants | 0 | 0

4. Primary Outcome: Number of Participants With a Clinical Laboratory Abnormality Leading to an AE
Description: Laboratory parameters included hematology (hematocrit, hemoglobin, red blood cell count, white blood cell count with differential [neutrophils, lymphocytes, monocytes, eosinophils, basophils], and platelet count); serum chemistries (blood urea nitrogen, creatinine, total bilirubin, aspartate aminotransferase, alanine aminotransferase, gamma-glutamyl transferase, alkaline phosphatase, total protein, sodium, potassium, bicarbonate, calcium, chloride, magnesium, inorganic phosphate, creatine kinase, lactate dehydrogenase, erythrocyte sedimentation rate, C-reactive protein, troponin, myoglobin, insulin-like growth factor 1, and cholesterol [(nonfasting]); urinalysis (color, pH, specific gravity, protein, glucose, ketones, and blood). Clinically significant laboratory abnormalities were based upon Investigator's discretion. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (up to Week 25)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - FSHD | Group B - LGMD2B and FSHD
Number analyzed (Participants) | 4 | 14
Participants | 0 | 4

5. Primary Outcome: Number of Participants With Vital Sign Abnormality Resulting in a TEAE
Description: The vital sign parameters that were evaluated included heart rate, systolic and diastolic blood pressure, and respiration rate as well as temperature. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (Up to Week 25)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - FSHD | Group B - LGMD2B and FSHD
Number analyzed (Participants) | 4 | 14
Participants | 0 | 3

6. Secondary Outcome: Percent Change From Baseline in Manual Muscle Testing (MMT) Score at Week 14
Description: MMT (muscle strength) was graded on a scale from 0 (no contraction palpable) to 5 (normal strength). Decreased muscle strength was indicated by a decreased score.
Time Frame: Baseline, Week 14
Population: Safety population included all participants who received at least 1 full or partial dose of ATYR1940 and had a post-infusion safety observation. Here, 'Overall Number of Participants Analyzed' (N) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Group A - FSHD | Group B - LGMD2B and FSHD
Number analyzed (Participants) | 4 | 13
percent change | -7.1 (13.38) | 4.3 (6.42)

ADVERSE EVENTS:
Time Frame: Up to End of Study (up to Week 25)
Description: Safety population included all participants who received at least 1 full or partial dose of ATYR1940 and had a post-infusion safety observation. Serious Adverse Event and Other Adverse Event data were prespecified to be collected by the participant's assigned arm, regardless of the participant's dose level.
Arm/Group | Group A - FSHD | Group B - LGMD2B and FSHD
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/14
Other Adverse Events (participants affected / at risk) | 4/4 | 14/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A - FSHD (N=4) | Group B - LGMD2B and FSHD (N=14)
Headache (Nervous system disorders) | 2 | 7
Presyncope (Nervous system disorders) | 0 | 2
Asthenia (General disorders) | 1 | 2
Fatigue (General disorders) | 2 | 1
Pyrexia (General disorders) | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Burning sensation (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Muscle contractions involuntary (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Feeling hot (General disorders) | 0 | 1
Infusion site pain (General disorders) | 0 | 1
Infusion site urticaria (General disorders) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Insulin-like growth factor increased (Investigations) | 0 | 1
Red blood cell sedimentation rate increased (Investigations) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2
Haematoma (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institutions and investigators agreed that no submission for publication or public disclosure will be made until after publication of the multi-center trial results by the sponsor, except in the following conditions:

* notification by sponsor that such multi-center trial submission is no longer planned;
* after the eighteen (18) month anniversary of the completion, abandonment or termination of such multi-center trial.